Protocol No. / Title: ZK-001/Safety and Pharmacokinetic Evaluation of Zika Virus Immune Globulin in Healthy

Volunteers (Protocol Version 3.1 June 5, 2018)

Site Code: Not applicable

Investigator:

TMF Section/Artifact name: 11.01.01 Statistical Analysis Plan

#### Details:

The purpose of this document is to outline any changes from the Statistical Analysis Plan (SAP) or important statistical analysis decisions that were made post-database lock and unblinding for study ZK-001.

The following issues are discussed:

- 1. Screen failure data
- 2. Pharmacokinetics (PK) neutralization assay deviation
- 3. PK analysis methodology

#### Assessm ent and Actions Taken:

- 1. Screen failure data were not collected in the clinical database for study ZK-001. These data were tracked by the site and shared with the Emergent clinical trial manager informally via an Excel tracker. At the end of the study, the screen failure data (total number of screen failures, 279, and associated reasons) were used in the Clinical Study Report (CSR) Section 12.1 text and Figure 2 subject disposition flow chart. It is acknowledged that these are unverified data.
- 2. A PK neutralization assay deviation is noted in APPENDIX I Documentation for Item #2 to this document. Briefly, the 1 hour, 3 hour and 8 hour time point concentrations for subject ZK-001-01-197 were incorrectly deemed a failed assay and repeated. The repeat data were used in the PK analysis rather than the original data; this anomaly is included in the PK Contributing Scientist report.
- 3. A number of changes were made to the ZK-001 PK analysis, some as a result of recommendations made by Nuventra Pharma Sciences in order to align our noncompartmental analysis (NCA) methodology to that of the industry standard Phoenix WinNonLin (Certara) software, as noted below.
  - The SAP states that, "All PK analyses include placebo subjects as well as ZIKV-IG subjects due to background antibody levels." When the PK concentration data were received, it was noted that the placebo subjects' values were all less than the lower limit of quantitation (LLOQ; 5 U/mL for binding assays and 15 U/mL for neutralization assay). This result was due to a background subtraction step applied during the assay. Consequently, PK analyses could not be performed for placebo subjects.
  - Imputation for PK analyses followed a PHUSE white paper Sections 6.2.1 and 6.2.2 to determine the following conventions:
     (https://www.phusewiki.org/wiki/images/e/ed/PhUSE\_CSS\_WhitePaper\_PK\_final\_25March2014.pdf)
    - o Predose values <LLOQ were set to zero and included in PK analyses.
    - $\circ$  Values prior to  $C_{max}$  (i.e., Day 1, 1 hour and 3 hour time points) and

Emergent BioSolutions, Inc. Printed on YYYY.MM.DD

CM224.01 Effective: 2018.Apr.12




# 'gent SAP Amendment 2 / Note to File

- <LLOQ were set to zero and included in PK analyses.</p>
- Values at the end of the curve <LLOQ were set to missing and excluded from PK analyses.
- PK concentrations for the anti-E protein binding assay included one value greater than the ULOQ of 300 U/mL. This value occurred at the Day 1, 1 hour time point for subject ZK-001-01-049. In the PK analysis, the value was imputed as 1.01 \* ULOQ or 303 U/mL and included in PK analysis.
- The SAP states that the "linear trapezoidal method" is used for PK analyses.
   In fact, the linear trapezoidal method was used for consecutive time points with level or increasing concentrations and the log-linear trapezoidal method was used for consecutive time points with decreasing concentrations per Nuventra recommendation.
- The terminal elimination constant lambda z was calculated using Intransformed data post-C<sub>max</sub> with a minimum of the last 3 points; more points were added and the adjusted r<sup>2</sup> was used to find the best model (except the second-best model was used if the difference in adjusted r<sup>2</sup> was <0.0001 and the second-best model used more data points, following <a href="https://www.lexjansen.com/pharmasug/2005/StatisticsPharmacokinetics/sp07.pdf">https://www.lexjansen.com/pharmasug/2005/StatisticsPharmacokinetics/sp07.pdf</a>). C<sub>max</sub> was excluded from the linear regression for lambda z calculation per Nuventra advice. No lower bound was placed on the adjusted r<sup>2</sup> value (such as 0.8 or 0.75) as Nuventra proposed.
- Additional PK parameters not mentioned in the SAP were reported per Nuventra recommendation: AUC%extrapolated, adjusted r² value, number of points used in lambda z calculation, and lower and upper range of times for points used in lambda z calculation for each subject.
   Additionally per Nuventra suggestion, geometric mean and geometric percent coefficient of variation were not displayed for ordinal time variables including t<sub>max</sub> and lower and upper limit of times for points used for lambda z.
- One subject, ZK-001-01-127, was removed from PK analyses as an outlier.
   This subject had a much later and lower C<sub>max</sub> value with an apparent absorption phase present. It is hypothesized that the subject received drug administration that inadvertently missed the vein and was injected intramuscularly; this hypothesis is supported by the adverse event of tissue swelling at the injection site.
- The PK concentration tables for each assay (Tables 14.3.6.1-3) were modified by excluding placebo subjects and removing the change from predose column (since individual background subtraction was performed as part of the assay). In addition, a column was added for the PK population with subject ZK-001-01-127 removed to permit comparison of the concentrations with and without this outlying subject.

CM224.01

Effective: 2018.Apr.12 



# emergent SAP Amendment 2 / Note to File

The PK parameter tables for each assay (Tables 14.3.7.1-3) were modified by adding a column for the PK population with subject ZK-001-01-127 removed to permit comparison of the parameters with and without this outlying subject. PK listings were not changed.

The PK profile figures for each assay (Figures 14.4.2.1-3) were modified by excluding subject ZK-001-01-127.

The individual PK profile Figure 14.4.2.4 was modified to overlay all three assays on the same plot for each subject; subject ZK-001-01-127 was retained.

The SAP states that, "values reported as below the limit of detection (LOD) are substituted with LOD/2." This rule was followed relative to the LLOQ (5 U/mL for binding assays and 15 U/mL for neutralization assay) for calculation of summary statistics, but not for PK analyses.

| Completed by: (Name, role) | Lead Biostatistician |
|----------------------------|----------------------|
| Signature: | Date: |

CM224.01

Effective: 2018.Apr.12  Protocol No. / Title: ZK-001/Safety and Pharmacokinetic Evaluation of Zika Virus Immune Globulin in Healthy Volunteers (Protocol Version 3.1 June 5, 2018)

Site Code: Not applicable

Investigator:

TMF Section/Artifact name: 11.01.01 Statistical Analysis Plan

#### Details:

According to the ZK-001 protocol and SAP, subjects with "a suitably low level of baseline anti-ZIKV E-protein binding antibodies" are to be included in the PK analysis population. Additionally, SAP (v1.0 18-APR-2019 Section 3.2 Analysis Populations) states "Subjects who exceed a threshold level of baseline anti-ZIKV E protein binding antibodies, to be determined after database lock, may be excluded from PK analysis." This statement was based on the erroneous assumption that all PK concentrations would be blinded; in fact, screening and baseline data were unblinded.

Consequently, the team decide to set the cutoff limit of baseline anti-ZIKV E-protein binding antibodies for inclusion in the PK population **prior** to database lock and examination of the blinded post-baseline PK data.

#### Assessment:

BIAD stated that the screening limit of 9.1 U/mL for anti-ZIKV E-protein binding antibodies was conservative and, following validation, could be confidently increased to 15-20 U/mL without affecting data integrity.

The screening and baseline antibody concentrations indicated that most subjects had low background anti-ZIKV E-protein binding antibody levels, with the maximum being 11.5 U/mL.

This SAP amendment 1/NTF was created to establish a baseline cutoff of 12 U/mL anti-ZIKV E-protein concentration for subject inclusion in the PK population. This document was prepared and signed off **prior** to database lock, and thus prior to examination of the blinded post-baseline PK data.

CM224.01

Effective: 2018.Apr.12 Page 1 of 2 Actions Taken:

- A limit of ≤12 U/mL baseline anti-ZIKV E-protein concentration was established for subject inclusion in the PK population. This was done prior to database lock.
- Application of this limit to current data indicates that no subject will be excluded from the PK analysis population due to high baseline antibody concentrations.
- See also TMF Section 12.8 NTF entitled "Threshold level of baseline anti-ZIKV E-protein binding antibodies" with the same date containing substantively the same information.

| Completed by: (Name, role) | Lead Biostatistician |
|----------------------------|----------------------|



# **Emergent BioSolutions STATISTICAL ANALYSIS PLAN**

# **Study Drug**

Zika Virus Immune Globulin (Human) (ZIKV-IG)

# **Protocol ZK-001**

# Safety and Pharmacokinetic Evaluation of Zika Virus Immune Globulin in Healthy Volunteers

| <b>Protocol Version</b> | Date |
|-------------------------|-------------|
| Protocol 1.0 | 30-OCT-2017 |
| Amendment 2.0 | 30-NOV-2017 |
| Amendment 2.1 | 10-JAN-2018 |
| Amendment 3.0 | 18-APR-2018 |
| Amendment 3.1 | 05-JUN-2018 |

**SAP Version** Date

**1.0 FINAL** 18-APR-2019



## SAP SIGNATURE PAGE

Signatures below indicate that the final version of the SAP or amended SAP is released for execution.

Study Statistician:

Biostatistician
Emergent BioSolutions

Signature / Date

Statistical Reviewer:

Sr. Manager, Biostatistics
Emergent BioSolutions

Signature / Date

Project Manager:

Clinical Project Manager
Emergent BioSolutions

Signature / Date



# TABLE OF CONTENTS

| TABLE | OF CONTENTS | 3 |
|---------|--------------------------------------|----|
| LIST OF | ABBREVIATIONS | 6 |
| 1. | INTRODUCTION | 8 |
| 2. | PROTOCOL SUMMARY | 8 |
| 2.1. | Study Objectives | 8 |
| 2.1.1. | Primary Objective | 8 |
| 2.1.2. | Secondary Objective | 8 |
| 2.2. | Study Design and Conduct | 8 |
| 2.3 | Study Endpoints | 9 |
| 2.3.1 | Efficacy Endpoints | 9 |
| 2.3.2 | Safety Endpoints | 9 |
| 2.3.2.1 | Primary Safety Endpoint | 9 |
| 2.3.2.2 | Secondary Safety Endpoints | 9 |
| 2.3.3 | Pharmacokinetic Endpoints | 9 |
| 2.4 | Power and Sample Size Considerations | 10 |
| 2.5 | Randomization and Blinding | 10 |
| 3 | DATA CONSIDERATIONS | 11 |
| 3.1 | Protocol Deviations | 11 |
| 3.2 | Analysis Populations | 11 |
| 3.3 | Multicenter Study | 11 |
| 3.4 | Analysis Time Points | 12 |
| 3.5 | Definition of Baseline | 12 |
| 3.6 | Treatment Groups | 12 |
| 3.7 | Coding Dictionaries | 12 |
| 4 | STATISTICAL ANALYSIS | 15 |
| 4.1 | Statistical Software | 15 |
| 4.2 | Summary Statistics | 15 |
| 4.3 | Derived Variables | 15 |
| 4.4 | Statistical Hypotheses | 16 |
| 4.5 | Handling of Missing Data | 17 |



| 4.6 | Adjustment for Covariates | 17 |
|--------|-------------------------------------------------|----|
| 4.7 | Subgroup Analysis | 17 |
| 4.8 | Multiplicity Adjustment | 17 |
| 5 | STUDY POPULATION CHARACTERISTICS | 17 |
| 5.1 | Subject Disposition | 17 |
| 5.2 | Protocol Deviations | 17 |
| 5.3 | Demographics and Other Baseline Characteristics | 17 |
| 5.3.1 | Demographics | 17 |
| 5.3.2 | Baseline Viral Markers | 18 |
| 5.3.3 | Medical History | 18 |
| 5.3.4 | Screening Smoking History | 18 |
| 5.3.5 | Breath Alcohol Test at Screening and Baseline | 18 |
| 5.3.6 | Urine Drug Test at Screening and Baseline | 18 |
| 5.3.7 | Pregnancy Test at Screening and Baseline | 18 |
| 5.3.8 | Screening Urinalysis | 18 |
| 5.3.9 | Screening Electrocardiogram | 19 |
| 5.3.10 | Concomitant Medications | 19 |
| 6 | EFFICACY ANALYSIS | 19 |
| 7 | SAFETY ANALYSIS | 19 |
| 7.1 | Extent of Exposure | 19 |
| 7.2 | Primary Safety Analysis | 19 |
| 7.2.1 | Adverse Events | 19 |
| 7.3 | Secondary Safety Analysis | 20 |
| 7.3.1 | Clinical Laboratory Tests | 20 |
| 7.3.2 | Viral Markers | 20 |
| 7.3.3 | Vital Signs | 20 |
| 7.3.4 | Physical Examinations | 21 |
| 7.4 | Pharmacokinetic Analyses | 21 |
| 7.4.1 | Anti-ZIKV E-protein Binding Antibodies | 21 |
| 7.4.2 | Anti-ZIKV NS1 Binding Antibodies | 22 |
| 7.4.3 | Anti-ZIKV Neutralizing Antibodies | 22 |

# Zika Virus Immune Globulin (Human) (ZIKV-IG) Protocol ZK-001



| 8 | SAFETY MONITORING COMMITTEE AND INTERIM ANALYSES | 22 |
|---|---|---|
| 8.1 | Safety Monitoring Committee | 22 |
| 8.2 | Interim Analyses | 22 |
| 9 | REFERENCES | 23 |
| 10 | APPENDIX I AESI PREFERRED TERM LIST | 24 |
| 10.1 | Preferred Terms for Modified Hypersensitivity SMQ | 24 |
| 10.2 | Preferred Terms for Modified Renal Dysfunction SMQ | 28 |
| 10.3 | Preferred Terms for Modified Aseptic Meningitis Syndrome SMQ | 29 |
| 10.4 | Preferred Terms for Modified Hemolysis SMQ | 29 |
| 10.5 | Preferred Terms for Modified Thrombosis SMQ | 30 |
| 10.6 | Preferred Terms for Modified Transfusion-related Acute Lung Injury SMO | 35 |



# LIST OF ABBREVIATIONS

| AE | Adverse event |
|---|---|
| AESI | Adverse event of special interest |
| AUC <sub>0-day 7</sub> | Area under the serum concentration curve from time 0 to day 7 |
| AUC <sub>0-inf</sub> | Area under the serum concentration curve from time 0 to infinity |
| AUC <sub>0-t</sub> | Area under the serum concentration curve from time 0 to the last measurable concentration |
| BMI | Body mass index |
| CL | Clearance |
| C <sub>max</sub> | Maximum observed concentration |
| CRF | Case report form |
| CRO | Contract research organization |
| CS | Clinically significant |
| CSR | Clinical study report |
| CTMS | Clinical trial management system |
| DENV | Dengue virus |
| ECG | Electrocardiogram |
| EDC | Electronic data capture |
| FSH | Follicle-stimulating hormone |
| HBV | Hepatitis B virus |
| HCV | Hepatitis C virus |
| HIV | Human immunodeficiency virus |
| IV | Intravenous |
| LOD | Limit of detection |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NAT | Nucleic acid testing |
| NCS | Not clinically significant |
| NS1 | Zika virus non-structural protein 1 |
| PD | Protocol deviation |
| PK | Pharmacokinetics |
| PR interval | Interval from the beginning of the P wave to the beginning of the Q wave |



| QA | Quality assurance |
|---|---|
| QRS duration | Duration from the beginning of the Q wave to the end of the S wave |
| QT interval | Interval from the beginning of the Q wave to the end of the T wave |
| QTcB interval | Bazett's correction of QT interval, $QT/(RR)^{1/2}$ , where RR is one cardiac cycle from the beginning of one R wave to the beginning of the next one |
| QTcF interval | Fridericia's correction QT interval, QT/(RR) <sup>1/3</sup> , where RR is one cardiac cycle from the beginning of one R wave to the beginning of the next one |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SDTM | Study Data Tabulation Model |
| SMC | Safety monitoring committee |
| SMQ | Standard MedDRA query |
| TLF | Tables, listings, and figures |
| T <sub>max</sub> | Time at which C <sub>max</sub> occurs |
| t <sub>1/2</sub> | Apparent first order terminal elimination half-life |
| $V_{\rm Z}$ | Volume of distribution following IV administration |
| WHO DD | World Health Organization Drug Dictionary |
| WNV | West Nile virus |
| ZIKV | Zika virus |
| ZIKV-IG | Anti-Zika Virus Immune Globulin (Human) |
| $\lambda_{\mathrm{z}}$ | Terminal elimination rate constant |



#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on Protocol ZK-001 "Safety and Pharmacokinetic Evaluation of Zika Virus Immune Globulin in Healthy Volunteers" (Version 3.1, 05JUN2018). This document specifies details of the definitions of the derived variables, analysis methods, assumptions and data handling conventions. The document is accompanied by mock-up tables, listings, and figures (TLF) shells. Some further details on the calculation of derived variables are provided as programmer's notes in the TLF shells. The TLF shells serve only as a guide for programming the final TLFs. They are working documents and can be updated as needed.

#### 2. PROTOCOL SUMMARY

# 2.1. Study Objectives

#### 2.1.1. Primary Objective

The primary objective of this study was to assess safety of Zika Virus Immune Globulin (ZIKV-IG) in healthy volunteers.

### 2.1.2. Secondary Objective

The secondary objective of this study was to determine pharmacokinetics (PK) of ZIKV-IG in healthy volunteers.

# 2.2. Study Design and Conduct

Study ZK-001 was a Phase 1, single-center, double-blind, randomized, placebo-controlled clinical trial to evaluate the safety and PK of ZIKV-IG in healthy non-pregnant volunteer subjects between the ages of 18 to 55 years with blood type O<sup>+</sup> or O<sup>-</sup>.

Sample size for ZK-001 was 30 subjects randomized to receive either one dose level of ZIKV-IG (n=19) or placebo (n=11; normal saline), referred to as study medication or treatment.

Dosing of the first 6 eligible subjects was staggered over three days, wherein 2 subjects per day were randomized 1:1 and dosed at least 3 hours apart with ZIKV-IG or placebo. The remaining subjects were randomized 2:1 in 4 cohorts of size 6 subjects. The protocol states that cohorts 2 through 5 were each to be dosed on a single day. However, scheduling constraints resulted in dosing of cohorts 2, 3 and 4 subjects spread over 3 days each (see Section 4.3 definition of cohort). A Safety Monitoring Committee (SMC) was convened after cohort 2 to review safety data through 72 hours post-dosing for the first 12 dosed subjects.

On Day 1, subjects received intravenous (IV) administration of either 50 mL of ZIKV-IG or 50 mL of placebo. The administered dose of ZIKV-IG was planned to be 4650 mg (93 mg/mL \* 50 mL).

Each subject was to be followed-up for 85 calendar days post-study treatment administration for safety (adverse events [AEs], laboratory tests, viral markers, vital signs and physical examinations) and pharmacokinetic assessments.



# 2.3 Study Endpoints

### 2.3.1 Efficacy Endpoints

There are no efficacy endpoints for this study.

#### 2.3.2 Safety Endpoints

#### 2.3.2.1 Primary Safety Endpoint

The primary safety endpoint is the number and severity of AEs.

#### 2.3.2.2 Secondary Safety Endpoints

Safety is evaluated based on the following endpoints:

- Adverse events
- Laboratory test results (hematology, blood chemistry)
- Viral markers (human immunodeficiency virus 1 and 2 [HIV], hepatitis B and C virus [HBV, HCV], Zika virus [ZIKV] IgM/IgG and nucleic acid testing [NAT] in serum and urine)
- Vital signs
- Physical examinations

### 2.3.3 Pharmacokinetic Endpoints

Primary PK analysis is based on the validated MagPix anti-ZIKV E-protein binding assay serum antibody concentrations. Analysis parameters include:

- AUC<sub>0-t</sub>: area under the concentration-time curve from time 0 to the last quantifiable concentration
- AUC<sub>0-day 7</sub>: area under the serum concentration curve from time 0 to day 7
- AUC<sub>0-inf</sub>: AUC<sub>0-t</sub> plus the additional area extrapolated to infinity
- C<sub>max</sub>: maximum observed concentration
- T<sub>max</sub>: time at which C<sub>max</sub> occurs
- $\lambda_z$ : terminal elimination rate constant
- $t_{1/2}$ : apparent first order terminal elimination half-life
- CL: total body clearance following IV administration
- V<sub>z</sub>: volume of distribution following IV administration

PK parameters are calculated using non-compartmental analysis (see Section 7.4).

In addition, results from a second, unvalidated binding assay are investigational only. This assay measures serum concentrations of antibodies that bind recombinant Zika virus non-structural protein 1 (NS1). NS1-binding PK parameters may be calculated if data permit.

Finally, PK parameters derived from ZIKV neutralizing antibody concentrations are estimated as a secondary PK analysis. See Section 7.4 for further details.



# 2.4 Power and Sample Size Considerations

Sample size for ZK-001 was 30 healthy volunteers; subjects were randomized to receive either one dose level of ZIKV-IG (n=19) or placebo (n=11). While there was no formal sample size calculation as this was a Phase 1 clinical trial evaluating safety and PK of one dose level of ZIKV-IG, 19 subjects treated with the study medication allows for safety evaluation and for calculation of PK parameters.

# 2.5 Randomization and Blinding

Subjects were randomized by cohort, except that the first 6 subjects (cohort 1A, 1B and 1C) were randomized 1:1 in pairs dosed at least 3 hours apart on the same day over the course of 3 days. The remaining subjects were randomized 2:1 in 4 cohorts of size 6 subjects. The protocol states that cohorts 2 through 5 were each to be dosed on a single day. However, scheduling constraints resulted in dosing of cohorts 2, 3 and 4 subjects spread over 3 days each (see Section 4.3 definition of cohort).

The contract research organization's (CRO) unblinded statistician created the final randomization schedule. A paper copy was shared with unblinded pharmacists at the CRO's Phase 1 clinical site for dispensation. Other unblinded personnel included subcontracted unblinded clinical trial monitors and a segregated sponsor unblinded medical monitor (who subsequently joined the sponsor company during the course of the trial). The segregated sponsor unblinded medical monitor served on the SMC (see Section 8.1). In addition, designated personnel at the sponsor's bioanalytical laboratory assigned to perform PK sample testing were unblinded, but PK data were stored in a protected server location. All other sponsor and CRO personnel involved in the conduct of the trial remained blinded until database lock and unblinding.

Access to information in the Medidata RAVE electronic data capture (EDC) system was blinded using role-based permissions. Randomization group and study treatment dispensing data were integrated with the clinical database prior to database lock, but unblinding data were removed from blinded data extracts by the CRO until after database lock to ensure maintenance of the blind. Study treatment dosing data were reconciled with the randomized treatment group for each subject by the unblinded monitors, and any deviations were reported in a separate repository from the blinded EDC.

Data external to the EDC included safety laboratory test results and PK concentration data. Laboratory data were converted to Study Data Tabulation Model (SDTM) datasets and were not considered unblinding. PK concentration data, considered unblinding, were retained by the sponsor's bioanalytical laboratory until after database lock and unblinding, when they were converted to SDTM for analysis and inclusion in the Clinical Study Report (CSR).



#### 3 DATA CONSIDERATIONS

#### 3.1 Protocol Deviations

Protocol deviations (PDs) were documented by the monitors and captured directly in the EDC; there were no unblinding PDs. There is no Clinical Trial Management System (CTMS) for the ZK-001 study.

PDs were graded as minor, major or critical. Minor PDs are defined as those that do not impact subject safety or the statistical analysis. Major PDs are those that potentially affect subject safety or the quality of the data evaluation. Critical PDs are those that do affect a subject's rights or safety or the quality of the data evaluation, or that show a pattern indicating intentional unauthorized deviation or fraud. PDs were categorized as follows:

- Missed procedures/assessments
- Procedures/assessments outside protocol window
- Order of procedures/assessments
- Missed visit
- Visit outside protocol window
- Inclusion/exclusion
- Randomization
- Informed consent
- Study drug administration
- Documentation
- Study restrictions
- Other

# 3.2 Analysis Populations

<u>Safety Population</u>: The safety population includes all subjects who receive any amount of study medication (ZIKV-IGIV or placebo) per the clinical database. In the case of incorrect treatment administration, subjects are analyzed according to the treatment received. The safety population is the primary analysis population for all non-PK analyses.

<u>PK Population</u>: The PK population includes subjects who have adequate PK data for analysis (a pre-dose sample and at least one measurable post-dose sample), are ZIKV-negative by NAT and serology testing and have a suitably low level of baseline anti-ZIKV E-protein binding antibodies. Subjects who exceed a threshold level of baseline anti-ZIKV E-protein binding antibodies, to be determined after database lock, may be excluded from PK analysis. Subjects are analyzed according to the treatment received.

# 3.3 Multicenter Study

This study was conducted at a single Phase 1 clinical center, located in Toronto, Ontario, Canada.



# 3.4 Analysis Time Points

Scheduled visits and assessment time points in the study include the following (see Table 1):

- Screening
- Baseline
- Day 1-2 hr pre-dose, 1 hr pre-dose, 15 min after start of dosing, end of dosing and 1, 3 and 8 hr post-dosing
- Day 2 24 hr post-dosing
- Day 3 48 hr post-dosing
- Day 4 72 hr post-dosing
- Day 6 120 hr post-dosing
- Day 8 168 hr post-dosing
- Day 10 216 hr post-dosing
- Day 12 264 hr post-dosing
- Day 15 336 hr post-dosing
- Day 22 504 hr post-dosing
- Day 29 672 hr post-dosing
- Day 43 1008 hr post-dosing
- Day 57 1344 hr post-dosing
- Day 85 or early withdrawal 2016 hr post-dosing

Early withdrawal data is not windowed to a scheduled visit and may be summarized separately as its own visit in selected tabulations.

### 3.5 Definition of Baseline

Baseline data are defined as the latest data collected prior to study medication dosing (ZIKV-IGIV or placebo).

# 3.6 Treatment Groups

Tables are presented by treatment group: ZIKV-IG or placebo. A total column is included for selected tables.

# 3.7 Coding Dictionaries

Medical history and AEs are coded to system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary version 21.0.

Concomitant medications are coded to preferred drug name using World Health Organization Drug Dictionary (WHO-DD) version March 2018. Anatomic therapeutic class coding is not performed.



Table 1Schedule of Events

| | Screening | Baseline | | | | | Po | st Study T | Treatment | Administr | ation Visits | * | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (within<br>35 days of<br>Baseline) | (Day -1;<br>within<br>24 hrs of<br>Day 1) | Day 1<br>(Dosing<br>Day) | Day 2<br>(Discharge<br>Day) | Day 3 | Day 4 | Day 6 | Day 8 | Day<br>10 | Day 12 | Day 15 | Day<br>22 | Day<br>29 | Day<br>43 | Day<br>57 | Day 85<br>or<br>Early<br>Withdrawal |
| Informed consent | X | | | | | | | | | | | | | | | |
| Eligibility | X | X | | | | | | | | | | | | | | |
| Medical history | X | $X^1$ | | | | | | | | | | | | | | |
| Complete physical exam | $X^2$ | $X^2$ | | | | | | | | | | | | | | X |
| Study treatment administration | | | X | | | | | | | | | | | | | |
| Vital signs <sup>3</sup> | X | X | $X^{4a}$ | X <sup>5</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| ECG | X | | | | | | | | | | | | | | | |
| Hematology | X | X | | X <sup>5</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Blood | X | X | | X <sup>5</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Urinalysis | X | | | | | | | | | | | | | | | |
| Drug (urine)<br>test | X | X | | | | | | | | | | | | | | |
| Alcohol<br>(breath) test | X | X | | | | | | | | | | | | | | |
| Pregnancy test | $X^6$ | $X^6$ | | | | | | | | | | | | | | X <sup>6</sup> |
| Viral markers | $X^7$ | X8 | | | | | | | | | | | | | | X <sup>9</sup> |
| PK sample collection | | | X <sup>4b</sup> | X <sup>5</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events | _ | | $X^{4b}$ | X <sup>5</sup> | X | X | X | X | X | X | X | X | X | X | X | X |



| | Screening Baseline | | · · | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (within<br>35 days of<br>Baseline) | (Day -1;<br>within<br>24 hrs of<br>Day 1) | Day 1<br>(Dosing<br>Day) | Day 2<br>(Discharge<br>Day) | Day 3 | Day 4 | Day 6 | Day 8 | Day<br>10 | Day 12 | Day 15 | Day<br>22 | Day<br>29 | Day<br>43 | <b>Day</b> 57 | Day 85<br>or<br>Early<br>Withdrawal |
| Concomitant medications | X | X | $X^{4b}$ | $X^5$ | X | X | X | X | X | X | X | X | X | X | X | X |

<sup>&</sup>lt;sup>1</sup> Update of medical history (if necessary).

NOTE: all study laboratory assessments will be performed by the Phase 1 clinic's reference laboratory, except for ZIKV IgG serology (screening and baseline samples) which will be performed by the sponsor's ZIKV IgG binding assay. The sponsor will evaluate subjects' PK samples with two in-house assays (a binding ZIKV antibody assay and a neutralizing ZIKV antibody assay).

<sup>&</sup>lt;sup>2</sup> Including assessment of BMI; height and body weight will be measured at Screening and only body weight again at Baseline.

<sup>&</sup>lt;sup>3</sup> Vital signs include temperature, sitting blood pressure, respiratory rate, pulse oximetry and pulse.

<sup>&</sup>lt;sup>4a</sup> Vital signs to be performed 2 hours (±15 min) and 1 hour (±15 min) prior to dosing, during the IV infusion at 15 minutes (±5 min) and at the end of the IV infusion (+5 min)], and post-dosing at 1 hour (±5 min), 3 hours (±30 min) and 8 hours (±1 hr).

<sup>&</sup>lt;sup>4b</sup> PK sample collection, adverse events and concomitant medications assessments at 1 hour (±5 min), 3 hours (±30 min) and 8 hours (±1 hr) post-dosing. Pre-dose (i.e., baseline) PK sample to be collected within 2 hours prior to dosing.

<sup>&</sup>lt;sup>5</sup> To be performed 24 hours (±3 hours) post-dosing.

<sup>&</sup>lt;sup>6</sup> At screening serum pregnancy test for female subjects of child-bearing potential and FSH assessment for post-menopausal female subjects. The serum pregnancy test is required only for women of childbearing potential for Baseline (Day -1) and Day 85 study visits.

<sup>&</sup>lt;sup>7</sup> Serology testing for HIV, HBV, HCV, DENV, WNV; ZIKV NAT (serum, urine) and ZIKV serology.

<sup>&</sup>lt;sup>8</sup> ZIKV NAT (serum, urine) and ZIKV serology testing.

<sup>&</sup>lt;sup>9</sup> Serology testing for HIV, HBV, HCV; ZIKV NAT (serum, urine) and ZIKV serology.

<sup>\*</sup> Day 1 includes 1 hour ( $\pm 5$  min), 3 hours ( $\pm 30$  min) and 8 hours ( $\pm 1$  hr) time-points **post-dosing**, Day 2 is 24 hours ( $\pm 3$  hrs), Day 3 is 48 hours ( $\pm 3$  hrs), Day 4 is 72 hours ( $\pm 3$  hrs), Day 6 is 120 hours ( $\pm 6$  hrs), Day 8 is 168 hours ( $\pm 6$  hrs), Day 10 is 216 hours ( $\pm 12$  hrs), Day 12 is 264 hours ( $\pm 12$  hrs), Day 15 is 336 hours ( $\pm 12$  hrs), Day 22 is 504 hours ( $\pm 12$  hrs), Day 29 is 672 hours ( $\pm 24$  hrs), Day 43 is 1008 hours ( $\pm 48$  hrs), Day 57 is 1344 hours ( $\pm 48$  hrs) and Day 85 is 2016 hours ( $\pm 72$  hrs) **post-dosing**.



#### 4 STATISTICAL ANALYSIS

#### 4.1 Statistical Software

Statistical analyses are implemented using SAS® v9.4 or higher.

# 4.2 Summary Statistics

Continuous endpoints are summarized by descriptive statistics including number of subjects, mean, standard deviation (SD), median, minimum and maximum. Categorical endpoints are summarized by the number of subjects, frequency and percentage. Precision is rounded to the number of decimal places in the original data, except mean and SD are rounded to one additional decimal place.

#### 4.3 Derived Variables

This section provides definitions of the derived variables. In some cases, the definitions are provided in the relevant sections.

**Age in years** is defined as integer part of ([date of informed consent – date of birth] / 365.25). If date of informed consent is missing or partial, then the screening visit date will be used.

**AEs of special interest (AESI)** is defined as a preferred term in the modified Standard MedDRA Query (SMQ) lists contained in Appendix I, Section 10. These include the following categories: hypersensitivity, acute renal dysfunction/failure, aseptic meningitis syndrome, hemolysis or hemolytic anemia, thrombotic events and transfusion-related acute lung injury.

**Analysis populations** (see Section 3.2)

**Body mass index (BMI)** is defined as weight (kg) divided by height squared (m<sup>2</sup>).

**Change from baseline** is defined as (value at post-baseline assessment – value at baseline). Percent change from baseline is defined as (change from baseline / value at baseline) \* 100.

**Cohort** is not collected in the case report form (CRF) but derived as follows based on randomization date and time:

- Cohort 1 comprises the first 6 subjects randomized. Two subjects per day dosed on 3 separate days are cohorts 1A, 1B and 1C, respectively (subjects 021 and 040 for 1A, 030 and 013 for 1B and 038 and 049 for 1C).
- Cohort 2 comprises the second 6 subjects randomized. Two subjects per day were dosed on 3 separate days (subjects 080 and 085 for 2A, 127 and 129 for 2B and 160 and 171 for 2C).
- Cohort 3 comprises the third 6 subjects randomized. One subject was dosed (subject 198 for 3A), then 3 subjects were dosed (subjects 197, 210 and 212 for 3B) and 2 subjects were dosed (subject 224 and 225 for 3C) on 3 separate days.



- Cohort 4 comprises the fourth 6 subjects randomized. Two subjects (subjects 226 and 232 for 4A) were dosed on the same day as the last 2 subjects in Cohort 3. Three subjects were dosed (subjects 088R, 231 and 240 for 4B) and one more subject was dosed (subject 249 for 4C) on 2 separate days.
- Cohort 5 comprises the last 6 subjects randomized. All 6 subjects were dosed on the same day as the last subject in Cohort 4 (subjects 273, 274, 277, 284, 001R and 309 for 5A).

**Completion** of study is defined as no primary reason for study discontinuation present on the end of study CRF page. The question, "Did the subject complete the study per protocol?" is not used because this question may be answered no for a completed subject with a PD.

**Concomitant medication** is defined as a medication that either starts before dosing and is ongoing at the study treatment dosing start time or a medication that starts during the study. If medication start or end date or start or end time is missing or partial, then any medication that could be concomitant is counted as concomitant.

**Duration of infusion** is defined as the difference between end time and start time of infusion (minus any interruption time) in minutes.

**Exposure, total** = defined as total volume (mL) administered.

**One month** = (365.25/12) days = 30.4375 days.

**PDs** (see Section 3.1)

**Study Day 1** is defined as the day of study treatment administration. The day prior to the study treatment infusion day is Day -1. There is no Day 0.

**Study day** = (assessment date - Day 1 date + 1) if the assessment is on or after the date of study drug administration. Study day = (assessment date - Day 1 date) if the assessment is before the date of study drug administration.

**Study medication or study treatment** = ZIKV-IG or placebo.

**Treatment, actual** is defined as the actual treatment given field on the study drug administration CRF.

**Treatment-emergent AE** = not defined for this study because AEs are collected only during or after study drug administration (i.e., all AEs are treatment-emergent).

**Treatment, randomized** is defined as the treatment assigned to the subject on the randomization schedule.

# 4.4 Statistical Hypotheses

Study ZK-001 was designed to assess safety of ZIKV-IG in healthy volunteers by examining the number and severity of AEs. No statistical hypotheses are tested for AE and serious AE (SAE) data.



# 4.5 Handling of Missing Data

For PK and laboratory data, values reported as below the limit of detection (LOD) are substituted with LOD/2; values reported as ">xx" or "<xx" are substituted with xx.

No other imputation rules are used, and no dates are imputed.

### 4.6 Adjustment for Covariates

Not applicable because no formal hypothesis is being tested.

### 4.7 Subgroup Analysis

For AE and SAE incidences, no formal subgroup analyses is performed.

# 4.8 Multiplicity Adjustment

Not applicable due to no formal hypothesis tests being conducted.

#### 5 STUDY POPULATION CHARACTERISTICS

### 5.1 Subject Disposition

Subject disposition, including early withdrawal reasons, are summarized and presented by treatment group for all randomized subjects. Tabulations include number of subjects randomized to the treatment, number of subjects who discontinued prior to study treatment administration and the reasons for early withdrawal and number of subjects who discontinued prior to completion of all study visits and the reasons for early withdrawal. Disposition data are listed by subject. In addition, subject membership in each analysis population is tabulated by treatment group as well as listed for the safety population. A disposition flow chart is provided.

#### **5.2 Protocol Deviations**

All PDs defined in Section 3.1 are presented by treatment group for the safety population. All PDs are listed.

# 5.3 Demographics and Other Baseline Characteristics

#### 5.3.1 Demographics

Demographic variables include: age (see definition in Section 4.3), sex, whether or not subject is female of child-bearing potential, race and ethnicity, height, baseline weight, body mass index (BMI; see definition in Section 4.3) and blood type (O<sup>+</sup> or O<sup>-</sup>). These variables are summarized using descriptive statistics by treatment group for the safety population and are listed. Eligibility data is listed only.



#### **5.3.2** Baseline Viral Markers

Screening serology results for dengue virus (DENV) and West Nile virus (WNV) pass or fail, are reported along with baseline ZIKV NAT results for serum and urine and baseline ZIKV IgM and IgG serology results. These variables are summarized using descriptive statistics by treatment group for the safety population and are listed.

### **5.3.3** Medical History

Medical history is coded to system organ class and preferred term using MedDRA dictionary version 21.0 and is tabulated for each system organ class and preferred term using frequency counts by treatment group for the safety population. Each subject is counted once in each system organ class and preferred term even if multiple events in that category occurred for the subject. Medical history is listed.

### **5.3.4** Screening Smoking History

Smoking history is solicited from each subject at screening and includes whether the subject currently smokes. If the subject is a current smoker the type (cigarettes or e-cigarettes) is recorded as well as the number of units per day. Smoking history results are listed only.

#### 5.3.5 Breath Alcohol Test at Screening and Baseline

Breath alcohol test is performed for each subject at screening and baseline visits and includes if the test was performed, if not performed reason why and result of the test (positive or negative). Breath alcohol test results are listed only.

#### 5.3.6 Urine Drug Test at Screening and Baseline

Urine drug test is performed for each subject at screening and baseline visits and includes if the test was performed, if not performed reason why, test name (amphetamine, benzodiazepine, cannabinoids, cocaine, opiates, oxycodone) and result of the test (positive or negative). Urine drug screen results are listed only.

#### 5.3.7 Pregnancy Test at Screening and Baseline

Serum pregnancy test and follicle stimulating hormone (FSH) results at screening and baseline visits for female subjects of child-bearing potential are listed only.

#### 5.3.8 Screening Urinalysis

Clinical laboratory tests for urine are performed at screening. Parameters to be tested include red blood cells, white blood cells, blood, bacteria, specific gravity, pH, glucose, bilirubin, urobilinogen, ketones, protein, nitrite, leukocyte esterase and squamous epithelial cells.

Assessments include whether a urine sample was collected, if not reason why, and the investigator's interpretation of these parameters as clinically significant or not clinically significant. Urinalysis results are listed only.



### 5.3.9 Screening Electrocardiogram

Electrocardiogram (ECG) test including ventricular rate, PR interval, QRS duration, QT interval, QTcF interval, and QTcB interval (see List of ) is performed at screening. Assessments include whether the test was performed, if not reason why and the investigator's interpretation of these parameters as normal, abnormal but not clinically significant, or abnormal and clinically significant. ECG test results are listed only.

#### 5.3.10 Concomitant Medications

Concomitant medications are coded to preferred drug name using WHO-DD March 2018. Concomitant medications are tabulated for the safety population by preferred drug name and by treatment group.

#### 6 EFFICACY ANALYSIS

There is no efficacy analysis for this study.

#### 7 SAFETY ANALYSIS

# 7.1 Extent of Exposure

The following study treatment (ZIKV-IG or placebo) infusion variables are summarized by treatment group for the safety population:

- Was study drug administered (yes or no)?
- Status of infusion (complete or incomplete).
- Was infusion interrupted (yes or no)?
- Total volume infused (mL).
- Duration of infusion (min).
- Randomized treatment (ZIKV-IG or placebo).

Study drug administration data are listed.

Treatment compliance is not applicable to this study since the investigational treatment is administered as a single dose only in the clinic on Day 1.

# 7.2 Primary Safety Analysis

#### 7.2.1 Adverse Events

AEs are coded to system organ class and preferred term using MedDRA dictionary version 21.0. AEs are summarized by treatment group for the safety population, including the following AE summary tables:

• AEs by system organ class and preferred term (includes serious and nonserious AEs)



- AEs by system organ class, preferred term, and maximum severity (includes serious and nonserious AEs)
- Treatment-related AEs by system organ class and preferred term (includes serious and nonserious AEs)
- Serious AEs
- Treatment-related serious AEs by system organ class and preferred term
- AEs of special interest (see definition in Section 4.3)

Each subject is counted once in each system organ class and preferred term even if multiple events in that category occurred for the subject. Assessment of causality is reported in the EDC as related or not related/no relationship. AEs where the causality assessment is missing after querying are excluded from summaries by relationship to study treatment. Assessment of severity is collected in the EDC as mild, moderate or severe. AEs with missing severity assessment after querying are excluded from summaries by severity.

### 7.3 Secondary Safety Analysis

### 7.3.1 Clinical Laboratory Tests

Laboratory values for hematology include white blood cell count, neutrophils, lymphocytes, monocytes, eosinophils, basophils, neutrophils, blood smear (morphology: platelets, red blood cells, white blood cells), hemoglobin, hematocrit, red blood cells, and platelets. Laboratory values for blood chemistry include glucose, urea, calcium, albumin, total bilirubin, sodium, potassium, chloride, alkaline phosphatase, lactate dehydrogenase (LD), gamma-glutamyl transferase (CGT), aspartate aminotransferase (AST), alanine aminotransferase (ALT), thyroid stimulating hormone (TSH), creatinine.

At each scheduled visit, values and change from baseline to each scheduled visit are summarized by treatment group for the safety population using descriptive statistics. The number and percentage of study subjects with hematology values clinically significantly outside the normal range at any time on study are summarized. Clinical laboratory data are listed.

#### 7.3.2 Viral Markers

Viral marker testing including HIV serology, HBV HBsAg, HCV serology, DENV serology, WNV serology, ZIKV NAT (serum, urine) and ZIKV serology (IgM and IgG) are performed at screening and at Day 85/ early withdrawal. ZIKV NAT (serum, urine) and ZIKV IgM and IgG serology testing results are updated at baseline. The test result (pass/fail) is summarized using frequency counts by treatment group for the safety population at each visit. Viral marker results are listed.

# 7.3.3 Vital Signs

Vital signs data include sitting systolic blood pressure, sitting diastolic blood pressure, respiratory rate, pulse, oral temperature and pulse oximetry. The investigator's interpretation of these parameters as normal, abnormal but not clinically significant, or abnormal and clinically significant is also collected. Vital signs at each scheduled visit and time point and change from



baseline to each scheduled visit and time point are summarized by treatment group for the safety population using descriptive statistics. The number and percentage of study subjects with vital signs values assessed as clinically significantly abnormal at any time on study are summarized. Vital signs data are listed.

### 7.3.4 Physical Examinations

A complete physical examination including general appearance, eye, ear, nose, throat, head and neck, respiratory, cardiovascular, gastrointestinal, musculoskeletal, dermatological, peripheral vascular, lymphatic, neurological, and mental status is performed at screening, baseline and upon study completion/ early withdrawal. Assessments include the investigator's interpretation of these parameters as normal, abnormal but not clinically significant, or abnormal and clinically significant. Physical examination results are listed only.

# 7.4 Pharmacokinetic Analyses

PK analyses are based on serum concentrations of binding and neutralizing ZIKV antibodies as described in this section. All PK analyses include placebo subjects as well as ZIKV-IG subjects due to background antibody levels.

### 7.4.1 Anti-ZIKV E-protein Binding Antibodies

The primary binding assay is a validated MagPix assay targeting anti-ZIKV antibodies that bind a recombinant Zika virus glycoprotein (E-protein). PK analysis using data from this assay comprises the primary PK analysis.

Serum concentration versus time data are analyzed by standard non-compartmental methods (i.e., linear trapezoidal method). Actual times and not nominal times are used in the analysis, and concentrations below the LOD are imputed as half of this value. The following PK parameters are calculated using non-compartmental analysis:

- AUC<sub>0-t</sub>: area under the concentration-time curve from time 0 to the last quantifiable concentration
- AUC<sub>0-day 7</sub>: area under the serum concentration curve from time 0 to day 7
- AUC<sub>0-inf</sub>: AUC<sub>0-t</sub> plus the additional area extrapolated to infinity
- C<sub>max</sub>: maximum observed concentration
- T<sub>max</sub>: time at which C<sub>max</sub> occurs
- $\lambda_z$ : terminal elimination rate constant
- $t_{1/2}$ : apparent first order terminal elimination half-life
- CL: total body clearance following IV administration
- V<sub>z</sub>: volume of distribution following IV administration

PK concentrations by visit and time point as well as calculated PK parameters are reported using descriptive statistics for the PK population by treatment group, including the placebo group, for E-protein binding antibodies. Serum concentration-time data are plotted by treatment group means ± standard deviation for E-protein binding antibodies, and individual subject profiles are provided. PK concentration and parameter data are listed.



# 7.4.2 Anti-ZIKV NS1 Binding Antibodies

An unvalidated, experimental MagPix binding assay measures serum concentrations of antibodies that bind to a recombinant Zika virus NS1 protein. PK analysis using data from this assay are investigational only. NS1-binding PK parameters may be calculated as described above if data permit.

# 7.4.3 Anti-ZIKV Neutralizing Antibodies

The neutralization assay is an xCelligence functional assay that assesses the ability of anti-ZIKV antibodies to kill the virus. PK analysis using data from this assay are considered secondary. PK parameters derived from ZIKV neutralizing antibody concentrations are estimated as described above.

#### 8 SAFETY MONITORING COMMITTEE AND INTERIM ANALYSES

### 8.1 Safety Monitoring Committee

An SMC consisting at a minimum of two blinded medical reviewers (Phase 1 clinic's medical monitor and sponsor's medical monitor) and one unblinded segregated medical monitor (who subsequently joined the sponsor company during the course of the trial) may recommend stopping the trial if the safety review identifies unforeseen adverse effects that impact subject safety.

The SMC process is further outlined in the Medical Monitoring Plan for this study. Strict procedures governing handling of unblinded data are in place to maintain the integrity of the study blind (see Section 2.5).

# 8.2 Interim Analyses

No interim analysis is planned.



# 9 REFERENCES

None.



# 10 APPENDIX I AESI PREFERRED TERM LIST

10.1 Preferred Terms for Modified Hypersensitivity SMQ

| 10.1 | Preferred Terms for Modified Hypersensi |
|-------|-----------------------------------------|
| Acute | e generalised exanthematous pustulosis |
| Admi | inistration related reaction |
| Admi | inistration site dermatitis |
| Admi | inistration site eczema |
| Admi | inistration site hypersensitivity |
| Admi | inistration site rash |
| Admi | inistration site urticaria |
| Aller | gic bronchitis |
| Aller | gic cough |
| Aller | gic eosinophilia |
| Aller | gic hepatitis |
| Aller | gic keratitis |
| Aller | gic myocarditis |
| Aller | gic oedema |
| Aller | gic otitis media |
| Aller | gic pharyngitis |
| Aller | gic reaction to excipient |
| Aller | gic respiratory disease |
| Aller | gic respiratory symptom |
| Aller | gic sinusitis |
| | gic transfusion reaction |
| | olitis allergic |
| Anap | hylactic reaction |
| Anap | hylactic shock |
| Anap | hylactic transfusion reaction |
| Anap | hylactoid reaction |
| Anap | hylactoid shock |
| Angio | pedema |
| | ritis allergic |
| Aspir | in-exacerbated respiratory disease |
| Atop | |
| | naritis allergic |
| | chospasm |
| | moral oedema |
| | unctival oedema |
| | unctivitis allergic |
| | eal oedema |
| | natitis |
| Derm | natitis acneiform |



| Dormatitic alloraic |
|-------------------------------------------------------|
| Dermatitis allergic |
| Dermatitis atopic |
| Dermatitis bullous |
| Dermatitis exfoliative |
| Dermatitis exfoliative generalised |
| Dermatitis psoriasiform |
| Drug eruption |
| Drug hypersensitivity |
| Drug reaction with eosinophilia and systemic symptoms |
| Eczema |
| Eczema nummular |
| Eczema vesicular |
| Eczema weeping |
| Encephalitis allergic |
| Encephalopathy allergic |
| Epidermal necrosis |
| Epidermolysis |
| Epidermolysis bullosa |
| Epiglottic oedema |
| Erythema multiforme |
| Erythema nodosum |
| Exfoliative rash |
| Eye allergy |
| Eye oedema |
| Eye swelling |
| Eyelid oedema |
| Face oedema |
| Fixed eruption |
| Giant papillary conjunctivitis |
| Gingival oedema |
| Gingival swelling |
| Gleich's syndrome |
| Haemorrhagic urticaria |
| Hand dermatitis |
| Henoch-Schonlein purpura |
| Henoch-Schonlein purpura nephritis |
| Hypersensitivity |
| Hypersensitivity myocarditis |
| Hypersensitivity vasculitis |
| Idiopathic urticaria |
| Immediate post-injection reaction |
| Immune-mediated adverse reaction |
| miniane mediated daverse reaction |



| Influsion related reaction |
|-------------------------------------------------|
| Infusion related reaction |
| Infusion site dermatitis |
| Infusion site eczema |
| Infusion site hypersensitivity |
| Infusion site rash |
| Infusion site recall reaction |
| Infusion site urticaria |
| Infusion site vasculitis |
| Injection related reaction |
| Injection site dermatitis |
| Injection site eczema |
| Injection site hypersensitivity |
| Injection site rash |
| Injection site recall reaction |
| Injection site urticaria |
| Injection site vasculitis |
| Interstitial granulomatous dermatitis |
| Intestinal angioedema |
| Kounis syndrome |
| Laryngeal oedema |
| Laryngitis allergic |
| Laryngospasm |
| Laryngotracheal oedema |
| Limbal swelling |
| Lip oedema |
| Lip swelling |
| Mouth swelling |
| Mucocutaneous rash |
| Multiple allergies |
| Nephritis allergic |
| Nodular rash |
| Oculomucocutaneous syndrome |
| Oculorespiratory syndrome |
| Oedema mouth |
| Oral allergy syndrome |
| Oropharyngeal blistering |
| Oropharyngeal oedema |
| Oropharyngeal spasm |
| Oropharyngeal swelling |
| Palatal oedema |
| Palatal swelling |
| Palisaded neutrophilic granulomatous dermatitis |



| Palpable purpura |
|------------------------------------------------------|
| Perioral dermatitis |
| Periorbital oedema |
| Pharyngeal oedema |
| Pruritus allergic |
| Rash |
| Rash erythematous |
| Rash follicular |
| Rash generalised |
| Rash macular |
| Rash maculo-papular |
| Rash maculovesicular |
| Rash morbilliform |
| Rash papulosquamous |
| Rash pruritic |
| Rash pustular |
| Rash rubelliform |
| Rash scarlatiniform |
| Rash vesicular |
| Reaction to excipient |
| Rhinitis allergic |
| Scleral oedema |
| Scleritis allergic |
| Scrotal oedema |
| Serum sickness |
| Serum sickness-like reaction |
| Skin necrosis |
| Skin reaction |
| Skin test positive |
| Stevens-Johnson syndrome |
| Swelling face |
| Swollen tongue |
| Symmetrical drug-related intertriginous and flexural |
| exanthema |
| Therapeutic product cross-reactivity |
| Tongue oedema |
| Toxic epidermal necrolysis |
| Toxic skin eruption |
| Tracheal oedema |
| Type I hypersensitivity |
| Type II hypersensitivity |
| Type III immune complex mediated reaction |



Type IV hypersensitivity reaction Urticaria Urticaria papular Urticaria pigmentosa Urticaria vesiculosa **Urticarial vasculitis** Vessel puncture site rash Vessel puncture site vesicles Asthma Asthma late onset Asthmatic crisis Auricular swelling Bronchial hyperreactivity Bronchial oedema Ear swelling Eosinophilic bronchitis Erythema Flushing Generalised erythema Generalised oedema Genital rash Genital swelling Haemolytic transfusion reaction Localised oedema Oedema mucosal Orbital oedema Penile oedema Penile swelling Perineal rash Pneumonitis Pruritus Pruritus generalised Respiratory tract oedema Scrotal swelling Seasonal allergy Skin swelling Sneezing Status asthmaticus Wheezing

# 10.2 Preferred Terms for Modified Renal Dysfunction SMQ

| Clamari | ılar vascular | dicardar |
|----------|---------------|----------|
| Gioinera | ılar vascular | uisoruei |



Hypertensive nephropathy Ischaemic nephropathy Malignant renal hypertension Nephroangiosclerosis Page kidney Renal aneurysm Renal arteriosclerosis Renal arteritis Renal artery arteriosclerosis Renal artery dissection Renal artery fibromuscular dysplasia Renal artery hyperplasia Renal artery occlusion Renal artery perforation Renal artery stenosis Renal artery thrombosis Renal embolism Renal hypertension Renal infarct Renal ischaemia Renal vascular thrombosis Renal vasculitis Renal vein embolism Renal vein occlusion Renal vein stenosis Renal vein thrombosis Renal vein varices Renal vessel disorder Renovascular hypertension Renal cortical necrosis Renal necrosis Renal papillary necrosis Renal tubular necrosis

# 10.3 Preferred Terms for Modified Aseptic Meningitis Syndrome SMQ

Meningitis aseptic

# 10.4 Preferred Terms for Modified Hemolysis SMQ

| Acute haemolytic transfusion reaction |
|---------------------------------------|
| Autoimmune haemolytic anaemia |
| Cold type haemolytic anaemia |
| Coombs direct test positive |



Coombs indirect test positive
Coombs negative haemolytic anaemia
Coombs positive haemolytic anaemia
Coombs test positive
Delayed haemolytic transfusion reaction
Extravascular haemolysis
Haemoglobin urine present
Haemoglobinaemia
Haemoglobinuria
Haemolytic anaemia
Haemolytic transfusion reaction
Haptoglobin decreased
Intravascular haemolysis
Warm type haemolytic anaemia

# 10.5 Preferred Terms for Modified Thrombosis SMQ

| Amaurosis |
|----------------------------------|
| Amaurosis fugax |
| Aortic thrombosis |
| Arterial occlusive disease |
| Arterial thrombosis |
| Basal ganglia infarction |
| Basilar artery occlusion |
| Basilar artery thrombosis |
| Blindness transient |
| Brachiocephalic artery occlusion |
| Carotid arterial embolus |
| Carotid artery occlusion |
| Carotid artery thrombosis |
| Cerebellar artery occlusion |
| Cerebellar artery thrombosis |
| Cerebral artery embolism |
| Cerebral artery occlusion |
| Cerebral artery thrombosis |
| Coronary artery embolism |
| Coronary artery occlusion |
| Coronary artery reocclusion |
| Coronary artery thrombosis |
| Embolism arterial |
| Femoral artery embolism |
| Hepatic artery embolism |



| Hepatic artery occlusion |
|---------------------------------------|
| Hepatic artery thrombosis |
| Iliac artery embolism |
| Iliac artery occlusion |
| Ischaemic cerebral infarction |
| Ischaemic stroke |
| Lacunar infarction |
| Leriche syndrome |
| Mesenteric arterial occlusion |
| Mesenteric arteriosclerosis |
| Mesenteric artery embolism |
| - |
| Myscardial infarction |
| Myocardial infarction |
| Myocardial necrosis |
| Papillary muscle infarction |
| Penile artery occlusion |
| Peripheral arterial occlusive disease |
| Peripheral arterial reocclusion |
| Peripheral artery occlusion |
| Peripheral artery thrombosis |
| Peripheral embolism |
| Popliteal artery entrapment syndrome |
| Post procedural myocardial infarction |
| Postinfarction angina |
| Precerebral artery occlusion |
| Precerebral artery thrombosis |
| Pulmonary artery occlusion |
| Pulmonary artery thrombosis |
| Renal artery occlusion |
| Renal artery thrombosis |
| Renal embolism |
| Retinal artery embolism |
| Retinal artery occlusion |
| Retinal artery thrombosis |
| Silent myocardial infarction |
| Spinal artery embolism |
| Spinal artery thrombosis |
| Splenic artery thrombosis |
| Splenic embolism |
| Subclavian artery embolism |
| Subclavian artery occlusion |
| Subclavian artery thrombosis |



| Superior mesenteric artery syndrome |
|----------------------------------------------------|
| Thrombotic microangiopathy |
| Thrombotic thrombocytopenic purpura |
| Transient ischaemic attack |
| Truncus coeliacus thrombosis |
| Vascular pseudoaneurysm thrombosis |
| Vertebral artery occlusion |
| Vertebral artery thrombosis |
| Axillary vein thrombosis |
| Brachiocephalic vein occlusion |
| Brachiocephalic vein thrombosis |
| Budd-Chiari syndrome |
| Cavernous sinus thrombosis |
| Cerebral venous thrombosis |
| Deep vein thrombosis |
| • |
| Deep vein thrombosis postoperative Embolism venous |
| Hepatic vein embolism |
| Hepatic vein occlusion |
| Hepatic vein thrombosis |
| Homans' sign positive |
| Iliac vein occlusion |
| Inferior vena cava syndrome |
| Inferior vena caval occlusion |
| Intracranial venous sinus thrombosis |
| Jugular vein occlusion |
| Jugular vein thrombosis |
| Mesenteric vein thrombosis |
| Mesenteric venous occlusion |
| Obstetrical pulmonary embolism |
| Obstructive shock |
| Ophthalmic vein thrombosis |
| Ovarian vein thrombosis |
| Pelvic venous thrombosis |
| Penile vein thrombosis |
| Portal vein occlusion |
| Portal vein thrombosis |
| Portosplenomesenteric venous thrombosis |
| Post procedural pulmonary embolism |
| Post thrombotic syndrome |
| Postoperative thrombosis |
| Postpartum venous thrombosis |



| Dulmonary embolism |
|------------------------------------|
| Pulmonary embolism |
| Pulmonary infarction |
| Pulmonary microemboli |
| Pulmonary thrombosis |
| Pulmonary vein occlusion |
| Pulmonary veno-occlusive disease |
| Pulmonary venous thrombosis |
| Renal vein embolism |
| Renal vein occlusion |
| Renal vein thrombosis |
| Retinal vein occlusion |
| Retinal vein thrombosis |
| Splenic vein occlusion |
| Splenic vein thrombosis |
| Subclavian vein occlusion |
| Subclavian vein thrombosis |
| Superior sagittal sinus thrombosis |
| Superior vena cava occlusion |
| Superior vena cava syndrome |
| Thrombosed varicose vein |
| Thrombosis corpora cavernosa |
| Transverse sinus thrombosis |
| Vena cava embolism |
| Vena cava thrombosis |
| Venoocclusive disease |
| Venoocclusive liver disease |
| Venous occlusion |
| Venous thrombosis |
| Venous thrombosis in pregnancy |
| Venous thrombosis limb |
| Visceral venous thrombosis |
| Administration site thrombosis |
| Adrenal thrombosis |
| Application site thrombosis |
| Arteriovenous fistula occlusion |
| Arteriovenous fistula thrombosis |
| Arteriovenous graft thrombosis |
| Atrial thrombosis |
| Basal ganglia stroke |
| Bone infarction |
| Brain stem embolism |
| Brain stem infarction |



| Brain stem stroke |
|-------------------------------------------------|
| Brain stem thrombosis |
| Cardiac ventricular thrombosis |
| Catheter site thrombosis |
| Cerebellar embolism |
| Cerebellar infarction |
| Cerebral infarction |
| Cerebral imarction |
| Cerebral nicroembolism |
| Cerebral microembolism Cerebral septic infarct |
| Cerebral thrombosis |
| Cerebral thombosis Cerebral vascular occlusion |
| Cerebrospinal thrombotic tamponade |
| Characteristics |
| Choroidal infarction |
| Coronary bypass thrombosis |
| Disseminated intravascular coagulation |
| Embolic cerebral infarction |
| Embolic pneumonia |
| Embolic stroke |
| Embolism |
| Graft thrombosis |
| Haemorrhagic adrenal infarction |
| Haemorrhagic cerebral infarction |
| Haemorrhagic infarction |
| Haemorrhagic stroke |
| Haemorrhagic transformation stroke |
| Haemorrhoids thrombosed |
| Heparin-induced thrombocytopenia |
| Hepatic infarction |
| Hepatic vascular thrombosis |
| Infarction |
| Infusion site thrombosis |
| Inner ear infarction |
| Intestinal infarction |
| Intracardiac thrombus |
| Mesenteric vascular occlusion |
| Microembolism |
| Optic nerve infarction |
| Pancreatic infarction |
| Paradoxical embolism |
| Paraneoplastic thrombosis |



| i . |
|-------------------------------------|
| Pituitary infarction |
| Placental infarction |
| Post procedural stroke |
| Postpartum thrombosis |
| Prosthetic cardiac valve thrombosis |
| Renal infarct |
| Renal vascular thrombosis |
| Retinal infarction |
| Retinal vascular thrombosis |
| Shunt occlusion |
| Shunt thrombosis |
| Spinal cord infarction |
| Splenic infarction |
| Splenic thrombosis |
| Stoma site thrombosis |
| Stroke in evolution |
| Testicular infarction |
| Thalamic infarction |
| Thromboangiitis obliterans |
| Thrombosis |
| Thrombosis mesenteric vessel |
| Thrombotic cerebral infarction |
| Thrombotic stroke |
| Thyroid infarction |
| Tumour embolism |
| Tumour thrombosis |

# 10.6 Preferred Terms for Modified Transfusion-related Acute Lung Injury SMQ

| Acute respiratory distress syndrome |
|---------------------------------------|
| Non-cardiogenic pulmonary oedema |
| Transfusion-related acute lung injury |
| Acute lung injury |